CLINICAL TRIAL: NCT04239274
Title: Spectral Correlates of Impulsivity in Patients With Traumatic Brain Injury: A Study of the Effect of Transcranial Electrical Stimulation of the Ventrolateral Prefrontal Cortex on Response Inhibition
Brief Title: Spectral Correlates of Impulsivity in Patients With Traumatic Brain Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled due to COVID
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Nathan Rowland, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00093356
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcranial Direct Current Stimulation (tDCS) (Experimental)
  Interventions: Device: transcranial direct current stimulation
- Transcranial Pulsed Stimulation tPCS (Experimental)
  Interventions: Device: transcranial pulsed current stimulation
- No Stimulation (Sham Comparator)
  Interventions: Device: Sham-no stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Subjects in this arm will receive one session of tDCS for 20 minutes at 2.0 milliamps.
  Arms: Transcranial Direct Current Stimulation (tDCS)
Device: transcranial pulsed current stimulation — Subjects in this arm will receive one session of tPCS for 20 minutes at 2.0 milliamps.
  Arms: Transcranial Pulsed Stimulation tPCS
Device: Sham-no stimulation — Subjects in this arm will receive one session of sham for 20 minutes.
  Arms: No Stimulation

SUMMARY:
Transcranial electrical stimulation (tES) is a non-invasive form of brain stimulation that has previously been to shown to have therapeutic potential in traumatic brain injury (TBI) patients. In this study, the study team will use a brain activity monitor (electroencephalogram, EEG) and a computer-based task to observe the effects of different forms of tES, like transcranial direct current stimulation (tDCS) and transcranial pulsed current stimulation (tPCS), on impulse control and sustained attention in people with TBI. Additionally, the study team will measure how much tDCS and tPCS affect the brain activity of a specific area of the brain associated with impulse control and attention. Problems with response inhibition have been shown to make rehabilitation more difficult for people with TBI. It also reduces social functioning and can also negatively affect job performance, which ultimately lead to a decreased quality of life. A better understanding of the effects of tES in TBI patients could be informative in finding out what its therapeutic potential is for this population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred to the PI for management of TBI
* Subject is at least 3 months post-injury at the time of consent
* Ages 25-70

Exclusion Criteria:

* Subjects with the inability to consent for themselves
* Subjects with body habitus that does not allow the EEG cap to be properly placed
* Presence of scalp injury or disease
* Allergic reaction to topical lidocaine jelly
* Prior intracranial surgery or skull-fracture over VLPFC
* Presence of hemorrhage on intracranial imaging
* Prior brain radiotherapy
* Prior history of intracranial tumor, intracranial infection, or cerebrovascular malformation
* Subjects with the inability to see and read from a computer screen
* History of any form of seizures prior to TBI or within 6 months of study participation
* Pregnancy

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Average Reaction Time During Stop Signal Task | Throughout study (1 hour)
  The Stop Signal Task (SST) is an assessment which requires participants to respond to various stimuli with a specific action and to not respond when a "stop" stimulus is presented.
EEG power in all frequency bands | Baseline and immediately post Stimulation
  They will be fitted with a standard EEG cap consisting of 32 EEG electrodes placed in the 10/20 international system format, a standardized system for EEG electrode placement. Frequency bands will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Rowland, MD,PhD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification may be shared as well as the study protocol, statistical analysis plan, and analytic code.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: For analyses to achieve aims in the approved proposal accessible by contacting the study principal investigator.